CLINICAL TRIAL: NCT02560272
Title: A Phase III, Double Blind, Parallel-controlled, Randomised Study to Evaluate the Safety and Immunogenicity of Haemophilus Influenzae Type b Conjugate Vaccine in Healthy Children 2 Months to 5 Years of Age
Brief Title: Safety and Immunogenicity of Haemophilus Influenzae Type b Conjugate Vaccine，Freeze-dried
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Minhai Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014L00216
Record Dates: First submitted 2015-09-19; First posted 2015-09-25 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Haemophilus Influenzae Type b Infections
Keywords: vaccine; haemophilus influenzae type b
MeSH Terms: conditions — Haemophilus Infections | interventions — Hiberix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minhai-HIB (Experimental): Participants at age 1 to 5 years of enrollment will receive one dose on Hib vaccine. Participants at age 6 to 11 months of enrollment will receive 2 doses on Hib vaccine at one months apart. Participants at age 2 to 5 months of enrollment will receive 3 doses on Hib vaccine at one months apart.
  Interventions: Biological: Minhai-HIB
- Act-HIB® (Active Comparator): Participants at age 1 to 5 years of enrollment will receive one dose on Hib vaccine. Participants at age 6 to 11 months of enrollment will receive 2 doses on Hib vaccine at one months apart. Participants at age 2 to 5 months of enrollment will receive 3 doses on Hib vaccine at one months apart.
  Interventions: Biological: Act-HIB®

INTERVENTIONS:
Biological: Minhai-HIB — 0.5ml, intramuscular
  Arms: Minhai-HIB
Biological: Act-HIB® — 0.5ml, intramuscular
  Arms: Act-HIB®

SUMMARY:
The study will evaluate the safety and immunogenicity of a haemophilus influenzae type b conjugate vaccine (Hib) in Healthy Children 2 Months to 5 Years of Age who have not been previously immunized with a Hib vaccine. Children 2 to 5 months of age will receive 3 doses of Hib vaccine, Children 6 to 11 months of age will receive 2 doses of Hib vaccine, Children 1 to 5 years of age will receive 1 dose of Hib vaccine, with each dose given approximately 1 month apart.

ELIGIBILITY:
Inclusion Criteria:

* Healthy permanent residence 2 months to 5 years old.
* Subjects who the investigator believes will comply with the requirements of the protocol should be enrolled in the study.
* Subjects and parent/guardian able to attend all scheduled visits and comply with all study procedures.
* Axillary temperature ≤37.0 ℃.

Exclusion Criteria:

* History of Haemophilus influenzae type b infection or vaccination of Haemophilus influenzae type b conjugate vaccine.
* Allergic history or any SAE after vaccination, such as allergy, urticaria, dyspnea, angioedema, celialgia.
* Receipt of blood or blood-derived products in the 3 months preceding vaccination
* Participation in another clinical study investigating a vaccine, drug in the 30 days preceding vaccination.
* Receipt of any live virus vaccine in the 15 days preceding vaccination.
* Receipt of any subunit vaccine and inactivated vaccine in the 7 days before vaccination.
* Febrile illness (temperature ≥ 38°C) in the 3 days or any acute illness/infection in the 7 days preceding vaccination.
* Thrombocytopenia.
* History of treatment for thyroid gland disease.
* Functional or anatomic asplenia.
* History of eclampsia, epilepsy, encephalopathy and mental disease or family disease.
* Any condition that, in the judgment of investigator, may affect trial assessment.

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1560 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects With Anti-polyribosylribitol Phosphate (Anti-PRP) Antibody Concentrations Greater Than or Equal to (≥) 0.15 Microgram Per Milliliter (µg/mL) and ≥ 1.0 µg/mL | 28 days after last dose of primary vaccination

SECONDARY OUTCOMES:
Number of Subjects With Any Solicited Local and General Symptoms | Within 7 days after any vaccination
Number of Subjects With Any Unsolicited Adverse Events (AEs) | Within 28 days after any vaccination
Anti-polyribosylribitol Phosphate (Anti-PRP) Antibody Concentrations | 28 days after last dose of primary vaccination

CONTACTS AND LOCATIONS:
Overall Officials: shengli xia, Principal Investigator — Henan Provincial Center for Disease Control and Prevention
Locations (1):
- Henan Provincial Center for Disease Control and Prevention, Zhengzhou, Henan, China